CLINICAL TRIAL: NCT03312920
Title: Investigating Memory Retrieval Improvement in Healthy Subjects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Planned changed based on the outcome of another study
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Sven Vanneste, Associate professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-132
Record Dates: First submitted 2017-10-12; First posted 2017-10-18 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Healthy Adults
Keywords: tDCS, accelerated learning, memory

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- active anodal tDCS (Experimental): active anodal tDCS with Face Name associate Memory task
  Interventions: Device: active anodal tDCS
- Sham tDCS (Sham Comparator): sham tDCS with Face Name associate Memory task
  Interventions: Device: sham tDCS
- active cathodal tDCS (Experimental): active cathodal tDCS with Face Name associate Memory task
  Interventions: Device: active cathodal tDCS

INTERVENTIONS:
Device: active anodal tDCS — active anodal tDCS with memory task
  Arms: active anodal tDCS
Device: sham tDCS — sham tDCS with memory task
  Arms: Sham tDCS
Device: active cathodal tDCS — active cathodal tDCS with memory task
  Arms: active cathodal tDCS

SUMMARY:
The purpose of this study is to investigate whether learning can be accelerated and associative memory performance improved in healthy subjects by applying transcranial Direct Current Stimulation (tDCS) during a Face Name memory task.

DETAILED DESCRIPTION:
Associative memory refers to remembering the association between two items, such as a face and a name or a word in English and the same word in another language. It is not only important for learning, but it is also one of the first aspects of memory performance that is impacted by aging and by Alzheimer׳s disease. For decades, neuroscientists have investigated associative learning and memory and ways to accelerate and enhance associative learning and memory.

Transcranial Direct Current stimulation (tDCS) is a non-invasive and painless electrical stimulation technique that has demonstrated to accelerate learning and improve memory in some studies. To investigate whether learning can be accelerated and associative memory improved by using tDCS, this study will compare the performance in a Face Name Associate memory task from 3 groups. The first group will get active aodal tDCS during the study phase of the Face Name Memory task, whereas the second group will get sham tDCS during the study phase of the task and the third group will get active cathodal tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years Native English Speaker

Exclusion Criteria:

* History of severe head injuries, epileptic insults, or heart disease. Severe psychiatric disorders and severe untreated medical problems. Contraindications for tDCS (pregnant women, implanted devices)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Associative Memory assessed by a Face Name Associate Memory experiment | Associate Memory is assessed after a 10 minutes break following the study phase
  Changes in performance in the Face Name Associate memory task is compared between the 2 groups (1. Real tDCS+ Face Name Associate memory task & 2. Sham tDCS+ Face Name Associate memory task) to investigate the influence of tDCS on Associative Memory.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- University of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No